CLINICAL TRIAL: NCT04902495
Title: Clinical and Radiographic Evaluation of Pulpotomies in Primary Molars Using Tricalcium Silicate Cements.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Francisco Guinot-Jimeno, Head of the pediatric dentistry department., Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UIC
Record Dates: First submitted 2020-06-30; First posted 2021-05-26 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Primary Molar Pulpotomy
MeSH Terms: interventions — tricalcium silicate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pulp Dressing MTA Angelus (Experimental): pulp therapy
  Interventions: Other: MTA HP Repair
- Pulp Dressing MTA Pro Root (Experimental): pulp therapy
  Interventions: Other: MTA Pro Root
- Pulp Dressing Biodentine (Experimental): pulp therapy
  Interventions: Other: Biodentine

INTERVENTIONS:
Other: MTA Pro Root — pulp therapy
  Arms: Pulp Dressing MTA Pro Root
Other: MTA HP Repair — pulp therapy
  Arms: Pulp Dressing MTA Angelus
Other: Biodentine — pulp therapy
  Arms: Pulp Dressing Biodentine

SUMMARY:
The objective of the study is to evaluate the success rate of pulpotomies in temporary molars using different types of hemostats and pulp coating materials based on tricalcium silicates, in patients who have attended the Dental Clinic of the International University of Catalonia (UIC).

DETAILED DESCRIPTION:
This prospective randomized clinical trial study has been approved by the

Scientific Committee in January of 2017 and by Ethics Committee (END-ECL- 2017-01) . It will be conducted in patients needing a vital pulp

therapy treatment at the Pediatric Dentistry Department of Universitat Internacional de Catalunya (Sant Cugat del Vallés, Barcelona, Spain). The necessary statistical sample size assuming an alpha risk of 0.05, a beta risk of 0.05 and a power of 95% sample, the required sample obtained by group resulted in 52. Given an estimate upwards of 20% of drop-outs in controls, the final size results in 62.4 (63 cases per group).

The data collection will be recollected using Excel program. Statgraphics Centurion XV software (StatPoint Technologies, Inc., Warrenton, VA, USA) will be used for statistical analysis. The chi-square test will be used and logistic regression analysis of the results will be performed to assess differences between groups with a significance level of P <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Responsible patients or parents or guardians who demonstrate that they understand the study and are willing to participate, as evidenced by signing the voluntary informed consent and receiving a signed and dated copy of the informed consent form.
* Children under 18 years of age with informed parental consent, correctly understood.
* Patient understands and is willing to comply with all study procedures and restrictions.
* Absence of clinical and radiographic evidence of pulp degeneration such as excessive bleeding, internal and / or external root resorption, destruction of the furcation.
* Asymptomatic and vital primary molars whose pulp exposure occurred during caries removal.

Exclusion Criteria:

* Patients with systemic pathologies (diabetes, inmunosuppresed or any clinically significant or relevant oral abnormality).
* Previous history of allergic reaction to local anesthesics or to the different constituents of the pulp agents to be studied.
* Pulp diagnosis of irreversible pulpits or pulp necrosis, root resorption, root fractures, pathological mobility, spontaneous pain, impossibility of restoration, and if pulpotomy is not the treatment of choice.

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 61 (Estimated)
Dates: Start 2017-01-12 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-12 (Estimated)

PRIMARY OUTCOMES:
visual examination | 12 months
  Clinical examination.Data will be recorded in terms of clinical signs of success.Clinical failure was determined by the subjective symptoms as explained by the participants and objective signs as recorded during clinical examination.
Radiographic Success | 12 months
  RX examination,Radiographic evaluation if success was performed according evidence of perirradicular or furcation pathosis or pathology root resorption.

SECONDARY OUTCOMES:
Radicular Radiolucency | 12 months
  RX examination,Radiographic evaluation if success was performed according evidence of perirradicular or furcation pathosis.
Internal Resorption | 12 months
  RX examination,Radiographic evaluation if success was performed according evidence of pathology root resorption.
External Resorption | 12 months
  RX examination,Radiographic evaluation if success was performed according evidence of pathology root resorption.
Furcation Radiolucency | 12 months
  RX examination,Radiographic evaluation if success was performed according evidence of perirradicular or furcation pathosis.
Symptoms of pain | 12 months
  Clinical examination,The patient will be recalled for control . Data will be recorded in terms of presence of symptoms, clinical and radiographic signs of success / failure, vertical and lateral percussion, periodontal probing and periapical and bitewing be implemented following the same methodology as in the initial evaluation.Clinical failure was determined by the subjective symptoms as explained by the participants.
Swelling | 12 months
  Clinical examination . Clinical failure was determined by the subjective symptoms as explained by the participants and objective signs as recorded during clinical examination including swelling.
Fistulation | 12 months
  Clinical and RX examination,The patient will be recalled for control .Clinical failure was determined by the subjective symptoms as explained by the participants and objective signs as recorded during clinical examination including abscess.
Pathological Mobility | 12 months
  Clinical examination,The patient will be recalled for control.Clinical failure was determined by the subjective symptoms as explained by the participants and objective signs as recorded during clinical examination including mobility.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat del Vallès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No